CLINICAL TRIAL: NCT05572814
Title: TRANSFORM3: Evaluation of Implementation Strategies of Teaching, Technology, and Teams to Optimize Medical Therapy in Cardiovascular Disease (T3)
Brief Title: Transform: Teaching, Technology, and Teams
Acronym: T3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American College of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 59648
Record Dates: First submitted 2022-09-27; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure; Type 2 Diabetes; Atrial Fibrillation
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Atrial Fibrillation | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Teaching - CardioSmart Resources + Clinician Education
- Decision Support (Active Comparator): Technology - Facilitated Solution (Existing Team)
  Interventions: Behavioral: Decision Support
- Referral (Active Comparator): Teams - Protocol-Supported Team, (Virtual GDMT Team)
  Interventions: Behavioral: Referral

INTERVENTIONS:
Behavioral: Decision Support — Prompts will be provided to clinicians signaling gaps in guideline-directed care
  Arms: Decision Support
Behavioral: Referral — Patients will be referred to an interdisciplinary, expert guideline-directed medical therapy team
  Arms: Referral

SUMMARY:
This initiative supports a quality improvement effort evaluating the use of strategies (including technology-based decision support, referral to a virtual GDMT team, and general educational tools/resources for clinicians and patients) to improve use of guideline-directed therapeutics known to lower cardiovascular (CV) events among patients with cardiovascular diseases of heart failure, atrial fibrillation and type 2 diabetes (T2D)/ASCVD with a specific focus on underserved populations and those with a history of health care disparities.

DETAILED DESCRIPTION:
TRANSFORM3 is a Quality Improvement initiative conducted in parallel to the current TRANSFORM CVRiD study and aligned with its goals of using a real-world population study to enable the American College of Cardiology Foundation ("ACCF") to better identify impactful ways to improve guideline directed medical therapy for patients. TRANSFORM3 is focused on improving GDMT use in underserved patients and patients with a history of health care disparities who have one or more of the following: heart failure, atrial fibrillation, and ASCVD/Type 2 diabetes.

There is a significant disconnect between increasing availability of effective and safe therapeutics that significantly reduce CV event risk in patients with Heart Failure, T2D and ASCVD, and Atrial Fibrillation-and clear guideline recommendations endorsing these therapies-but very low adoption in clinical practice with the majority of eligible patients that are most likely to benefit from these therapies not receiving them. A high proportion of patients have more than one of these conditions further reducing the chances of receiving optimal guideline directed medical therapy and avoiding the CV events they are designed to prevent.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years
2. Personal access to a computer and/or Smartphone for app download
3. Heart Failure (reduced and preserved ejection fraction) AND/OR
4. Atrial Fibrillation with CHA2DS2-VASc score greater than or equal to 2 in men and greater than or equal to 3 in women AND/OR
5. T2D and ASCVD, defined as follows:

   1. Known CAD, prior ACS, or coronary artery revascularization
   2. Prior TIA/stroke or known carotid or intracerebral atherosclerosis
   3. Prior PAD including requiring revascularization

Exclusion Criteria:

All patients

1. Current or anticipated participation in an interventional clinical trial of a drug/device
2. Currently receiving comfort care or enrolled in hospice
3. Life expectancy <1 year
4. Pregnancy or active breastfeeding
5. Current or anticipated participation in an interventional clinical trial (other than TRANSFORM3 GDMT)
6. Patients without a clinical encounter within three years of study start date

Heart Failure patients:

1. History of or plan for heart transplantation or left ventricular assist de-vice
2. Palliative chronic inotropic therapy
3. NYHA Class 4 heart failure

Atrial Fibrillation patients:

1. Current prescription for OAC
2. Reversible cause of atrial fibrillation, such as post-cardiothoracic surgery or thyrotoxicosis
3. History of ischemic stroke in prior 7 days
4. Transient ischemic attack in prior 3 days
5. Platelet count <70,000/ml
6. Hemoglobin concentration <8g/dl
7. History of or condition associated with increased bleeding risk, such as hemophilia
8. Major surgical procedure or trauma within 14 days
9. Clinically significant gastrointestinal bleeding within 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adoption of evidence-based CV-risk reduction and disease management therapies for HF, AF, and T2D/ASCVD. This data will be found in the patient's medical record. | 9 months
  GDMT baseline to 9 month change in average composite endpoint of receiving the main classes of drugs (50% or higher of target doses for HF) among eligible patients. We're aiming to see a change or increase in guideline-directed care where there was an original gap.

SECONDARY OUTCOMES:
Quality of Life Outcome-MMA-4 | Study duration up to 1 year.
  Difference in patient reported outcomes on Morisky Medication Adherence Scale (MMAS-4) from baseline, 3 and at 9 months.
Quality of Life Outcome-KCCQ-12 | Study duration up to 1 year.
  Difference in patient-reported outcome/KCCQ-12 scores from baseline to 9 months (applicable to HFrEF and HFpEF study cohorts only).
Quality of Life Outcome-PAM | Study duration up to 1 year.
  Difference in patient reported outcomes on Patient Activation Measure® (PAM) from baseline, 3 and at 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: James MD Januzzi, MD, Principal Investigator — Massachusetts General Hospital; Ankeet S Bhatt, MD, Principal Investigator — Kaiser Permanente; Andrew Oseran, MD, Principal Investigator — Massachusetts General Hospital; Megan Welch, MD, Principal Investigator — Massachusetts General Hospital; Jagmeet Singh, MD, Principal Investigator — Massachusetts General Hospital; Muthiah Vadduganathan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Cardiology Center of Amarillo, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT05572814/Prot_000.pdf
  • Informed Consent Form (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT05572814/ICF_001.pdf